CLINICAL TRIAL: NCT02299622
Title: Establishment of Personalized Cancer Medicine Using Samsung Cancer Sequencing Platform in Lung Cancer/Mediastinal Tumor/ Head & Neck/Esophageal Cancer/Rare Cancer (PerSeq: Personalized Sequence)
Brief Title: Personalized Sequence for Thoracic, Esophageal, and H&N Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Professor, Samsung Medical Center
Other Study IDs: 2013-10-112
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh tissue
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Genetic test — Next-generation sequencing (AmpliSeq) & fusion analysis

SUMMARY:
The next generation of personalized medical treatment according to the type of personal genetic information are evolving rapidly. The genome analysis needs systematic infra and database based on personal genetic information Therefore, a big data of genome-clinical information is important.

DETAILED DESCRIPTION:
To determine the feasibility of the use of tumor's molecular profiling and targeted therapies in the treatment of advanced cancer and to determine the clinical outcome(PFS, duration of response and overall survival) of patients with advanced cancer, the investigators are going to take a fresh tissue of patients and process molecular profiling.

ELIGIBILITY:
Inclusion Criteria:

* metastatic, histologically confirmed NSCLC, head & Neck Cancer, Esophageal cancer

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic, histologically confirmed NSCLC, head & Neck Cancer, Esophageal cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2022-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the spectrum of targetable genetic mutation in evaluated cancer specimens (for example, % of EGFR T790M mutation, BRAF mutation, or ALK mutation) | 3 years
  The pattern of the tumor's molecular profiling in advanced thoracic (lung, esophagus, or tthymic) cancer

CONTACTS AND LOCATIONS:
Overall Officials: Keunchil Park, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea